CLINICAL TRIAL: NCT05512728
Title: Efficacy of Virtual Reality Distraction Technique for Anxiety and Pain Control in Orthopedic Forearm Surgeries Performed Under Supraclavicular Brachial Plexus Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Haitham Hassan Eltrabily, lecturer of anasthesia and pain management, Cairo University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: MS-389-2020
Record Dates: First submitted 2022-08-20; First posted 2022-08-23 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Anesthesia
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: Categorical variables will be assessed using the chi-square or Fischer's exact test where appropriate. Normally distributed data will be presented as the mean (SD). Midazolam consumption and hemodynamic variables with a normal distribution will be analyzed using two-way analyses of variance with repeated measures and Dennett's post hoc test as appropriate. Data that are not normally distributed (by the Kolmogorov-Smirnov test) are presented as the median (range) and will be analyzed with the Kruskal-Wallis test as appropriate. The software SPSS v15.0 for Windows (SPSS, Inc, Chicago, IL, United States) will be used for statistical analysis
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- midazolam group (Placebo Comparator)
  Interventions: Drug: Midazolam
- VR group (Active Comparator)
  Interventions: Device: VR

INTERVENTIONS:
Device: VR — The IVR environment was provided by Shinecon VR (Shinecon, china). Shinecon VR features, have a large field of view and high-quality display; with aspheric lens , lens diameter 40MM, view angle 108 , sharpness 99%, visibility 100%, color .38MM and pupillary distance adjustment 65 MM.
  The shinecon VR setup was powered by a HUAWEI Y7 prime phone running the freely available IVR software.
  Shinecon VR provides videos for nature, forest, wind, desert and animals. That included noise-cancelling headphones playing background sound from the IVR simulation.
  Arms: VR group
Drug: Midazolam — • (titration of 0.05 mg/kg per dose) according to Modified Wilson sedation scale Score to achieve grade 1 (Oriented, eyes may be closed but can respond to 'Can you tell me your name?' 'Can you tell me where you are right now?'
  Arms: midazolam group

SUMMARY:
Invistigators hypothesized that using of VR distraction technique during performing peripheral regional anesthesia (supraclavicular block) would lead to better perioperative analgesia and less anxiety.

DETAILED DESCRIPTION:
Methodology I. Study design This is a controlled randomized prospective study. II. Study setting and location The study will be conducted at Cairo University Hospital - orthopedic surgery unit.

III. Study population Participants will be adult patients (above 18 years), ASA I-II, scheduled for elective forearm orthopedic surgeries under ultrasound guided supraclavicular approach for brachial plexus block.

IV. Study Procedures

1. Randomization Patients will be randomly allocated by a computer-generated table into one of the study groups; the randomization sequence will be concealed in sealed envelopes. Patients and data collector will be blind to group assignment.
2. Study Protocol Following approval from Ethics and Research Committee of Anesthesia Department, Faculty of Medicine, Cairo University, All patients will be subjected to systematic preoperative assessment including history taking, physical examination, and review of the results of routine investigations.

Upon arrival to the preparation room: A 20 gauge IV cannula is inserted into a peripheral vein then patients will be transferred to the operating room where basic monitoring Electrocardiography (ECG), Non-invasive Blood Pressure (NIBP) and pulse oximetry are attached. Baseline heart rate, blood pressure, oxygen saturation and respiratory rate will be recorded.

All patients will receive ultrasound guided supraclavicular block. The skin is disinfected and the transducer is positioned in the transverse plane immediately proximal to the clavicle, the transducer is tilted caudally, as if to image the chest contents, to obtain a cross-sectional view of the subclavian artery the brachial plexus is seen as a collection of hypo echoic oval structures posterior and superficial to the artery... Using a 25- to 27-gauge needle, 1-2 mL of local anesthetic is injected into the skin 1 cm lateral to the transducer .The distribution of local anesthetic via small-volume injections is observed as the needle advances through tissue layers (hydro-localization); small-volume injections are used to avoid inadvertent needle insertion into the brachial plexus. The block needle is then inserted in plane toward the brachial plexus, in a lateral-to-medial direction... Insertion of the needle into the sheath is often associated with a palpable "pop." After careful aspiration, 1-2 mL of local anesthetic is injected to confirm proper needle placement. When the injection displaces the brachial plexus away from the needle, an additional advancement of the needle 1-2 mm closer to the plexus may be required to accomplish adequate local anesthetic spread. When the injection of local anesthetic does not appear to result in a spread around the brachial plexus, needle repositioning may be necessary. Typically, 20-25 mL of local anesthetic is required for adequate block.

After local anesthetic injection through the block needle, measurements of brachial plexus blockade will be performed every 5 minutes until 30 minutes. Sensory blockade of the musculocutaneous, median, radial, and ulnar nerves was graded according to a 3-point scale using a cold test: 0 = no block, 1 = analgesia (patient can feel touch, not cold), 2 = anesthesia (patient cannot feel touch). Sensory blockade of the musculocutaneous, median, radial, and ulnar nerves will be assessed on the lateral aspect of the forearm, the volar aspect of the thumb, the lateral aspect of the dorsum of the hand, and the volar aspect of the fifth finger, respectively. Motor blockade will be also graded on a 3-point scale: 0 = no block, 1 = paresis, 2 = paralysis. Motor blockade of the musculocutaneous, radial, median, and ulnar nerves was evaluated by elbow flexion, thumb abduction, thumb opposition, and thumb adduction, respectively. Overall, the maximal composite score was 16 points. We will consider the patient ready for surgery when a minimal composite score of 14 points is achieved, provided the sensory block score is equal or superior to 7 of 8 points. (12) If, after 30 minutes, the composite score was <14 points, the patient will be excluded from the study and further management will be according to discretion of the attending anesthetist.

Patients in control group will not receive any additional management Patient in the VR group, before wearing the device, they will have the procedure explained to them, and reassured that they can terminate the VR session any time during the procedure. The VR set will be applied before performing the supraclavicular block and will be removed at the end of the procedure before leaving the operating room.

IVR simulation used:

The IVR environment was provided by Shinecon VR (Shinecon, china). Shinecon VR features, have a large field of view and high-quality display; with aspheric lens , lens diameter 40MM, view angle 108 , sharpness 99%, visibility 100%, color .38MM and pupillary distance adjustment 65 MM.

The shinecon VR setup was powered by a HUAWEI Y7 prime phone running the freely available IVR software.

Shinecon VR provides videos for nature, forest, wind, desert and animals. That included noise-cancelling headphones playing background sound from the IVR simulation.

•

Intraoperative sedation:

* (titration of 0.05 mg/kg per dose) according to Modified Wilson sedation scale Score to achieve grade 1 (Oriented, eyes may be closed but can respond to 'Can you tell me your name?' 'Can you tell me where you are right now?'
* titration of analgesia (fentanyl 1 mcg/kg per dose) according to numeric pain score to reach Zero pain.
* titration will be administered to all patients according to the attending anesthetist dissertation

Ultrasound-guided supraclavicular brachial plexus block simulating a single injection between the subclavian artery (SA) and the first rib Measured Parameter Demographic data of the patient

* Hemodynamics (heart rate, systolic and diastolic arterial blood pressure) will be recorded at baseline (upon patient admission to OR), 1 min after block then every 5 minutes till skin incision, 1 minute after skin incision and every 5 minutes till skin closure
* Total dos of midazolam needed for patient to relieve anxiety.
* The total dose of fentanyl
* The VR group, time required to set-up the virtual reality device, session lengths, early discontinuation, adverse events, such as: headache, nausea, or vomiting; and proportion of patients wishing to use the technology again
* The sedation level will be monitored using Modified Wilson sedation scale Score Description

  1. Oriented, eyes may be closed but can respond to 'Can you tell me your name?' 'Can you tell me where you are right now?'
  2. Drowsy; eyes may be closed, arousable only to command: '(name), please open your eyes'.
  3. Arousable to mild physical stimulation (earlobe tug)
  4. Unarousable to mild physical stimulation
* The pain level will be monitored using numeric pain scale

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II. patients scheduled for elective forearm orthopedic surgeries under ultrasound guided supraclavicular approach for brachial plexus block with good mental function.

Exclusion Criteria:

* Patient's refusal.

  * Known allergy to local anesthetics.
  * Bleeding disorders, Use of any anti-coagulants.
  * Inability to provide informed consent.
  * Patient with psychiatric disorders.
  * Sensory impairment (blindness, deafness).
  * Any technical problem preventing proper fitting of the glasses to the patient face
  * patients with cognitive impairment, epilepsy or with claustrophobia
  * patients with suspected eye infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-20 (Actual); Primary Completion 2022-12-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
● To estimate amount of IV sedation needed for the patient | (time from block needle entry till the end of the procedure)

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided